CLINICAL TRIAL: NCT02441972
Title: Phase 1 Study of 18F-Al-NOTA-PRGD2 in Cancer Diagnostics
Brief Title: Clinic Study of 18F-Al-NOTA-PRGD2 in Cancer Diagnostics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi No. 4 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LS2011051
Record Dates: First submitted 2015-04-21; First posted 2015-05-12 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2016-12

CONDITIONS: Tumors; Carcinoma, Bronchogenic; Breast Carcinoma; Cancer of Head and Neck; Lymphoma, Malignant; Soft Tissue Neoplasms
MeSH Terms: conditions — Neoplasms; Carcinoma, Bronchogenic; Breast Neoplasms; Head and Neck Neoplasms; Lymphoma; Soft Tissue Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-Al-NOTA-PRGD2 PET/CT (Experimental): Imaging with 18F-Al-NOTA-PRGD2 PET/CT.
  Interventions: Drug: 18F-Al-NOTA-PRGD2 PET/CT

INTERVENTIONS:
Drug: 18F-Al-NOTA-PRGD2 PET/CT — 18F-Al-NOTA-PRGD2(PET imaging agent) given by vein before PET scans.Perform PET/CT for each enrolled volunteer or patient at 60-90min.
  Other Names: 18F-Alfatide II PET/CT

SUMMARY:
The purpose of this study is to determine whether 18F-Al labeled RGD is safety and effective for cancer diagnosis and therapy response.

DETAILED DESCRIPTION:
Observe radiation dose to healthy volunteers and patients; the correlation between integrin level and tumor/metastases uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers or patients with age more than 18 yeas;
2. The patients have been diagnosed with cancer or suspected with cancer;
3. It must fulfill the ethical requirements and subjects have signed an informed consent.

Exclusion Criteria:

1. Pregnancy or nursing mothers;
2. Having drugs or alcohol dependence;
3. Hypersensitive to the active or inactive ingredients of the study drug;
4. Having attended other drug clinical trials within three months;
5. Cardiac functional insufficiency;
6. Hepatic and renal function insufficiency;
7. Hypertensive patients with serious complications;
8. Endangering the safety of life.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety data included vital signs (blood pressure, respiratory rate, heart rate, and body temperature) (composite) | 1 day
  Safety data were collected before and after injection of 18F-Al-NOTA-PRGD2. physical examination; ECG; laboratory parameters (blood routine, liver function and kidney function) and adverse events.

SECONDARY OUTCOMES:
radioactive distribution of normal organ, standard uptake value of tumor | 60 minutes
  Visual analysis whole body 18F-Al-NOTA-PRGD2 PET;Regions of interest (ROIs) were drawn manually on each image with the assistance of corresponding CT images. The results were expressed as standardized uptake value (SUV).
Diagnostic performance analysis to assess "sensitivity,specificity,accuracy,etc" | 1 day-1 year
  compare the Diagnostic outcome to pathology or clinic follow-up,then to gather statistics of sensitivity,specificity,accuracy,etc.

CONTACTS AND LOCATIONS:
Overall Officials: Weixing Wan, Professor, Study Chair — Wuxi No. 4 People's Hospital
Locations (1):
- Wuxi No. 4 People's Hospital, Wuxi, Jiangsu, China

REFERENCES:
- [Result] Beer AJ, Haubner R, Sarbia M, Goebel M, Luderschmidt S, Grosu AL, Schnell O, Niemeyer M, Kessler H, Wester HJ, Weber WA, Schwaiger M. Positron emission tomography using [18F]Galacto-RGD identifies the level of integrin alpha(v)beta3 expression in man. Clin Cancer Res. 2006 Jul 1;12(13):3942-9. doi: 10.1158/1078-0432.CCR-06-0266. PMID 16818691
- [Result] Beer AJ, Lorenzen S, Metz S, Herrmann K, Watzlowik P, Wester HJ, Peschel C, Lordick F, Schwaiger M. Comparison of integrin alphaVbeta3 expression and glucose metabolism in primary and metastatic lesions in cancer patients: a PET study using 18F-galacto-RGD and 18F-FDG. J Nucl Med. 2008 Jan;49(1):22-9. doi: 10.2967/jnumed.107.045864. Epub 2007 Dec 12. PMID 18077538
- [Derived] Wang L, Zhu X, Xue Y, Huang Z, Zou W, Zhang Z, Yu M, Pan D, Wang K. Ultrasensitive detection of uveal melanoma using [18F]AlF-NOTA-PRGD2 PET imaging. EJNMMI Res. 2024 Jul 5;14(1):62. doi: 10.1186/s13550-024-01123-4. PMID 38967722